CLINICAL TRIAL: NCT05888519
Title: Evaluation of Safety and Tolerability of Investigational Ocular Lubricants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DEP918-E001
Record Dates: First submitted 2023-05-09; First posted 2023-06-05 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FID123300/FID123301/FID122505 (Other): FID123300 ocular lubricant in Period 1, followed by FID12330 ocular lubricant in Period 2, followed by FID122505 ocular lubricant in Period 3, as randomized. For each period, the subject will receive one drop in each eye for one day. A 1-4 day washout will separate each period.
  Interventions: Other: FID123300 ocular lubricant; Other: FID123301 ocular lubricant; Other: FID122505 ocular lubricant
- FID123301/FID122505/FID123300 (Other): FID123301 ocular lubricant in Period 1, followed by FID122505 ocular lubricant in Period 2, followed by FID123300 ocular lubricant in Period 3, as randomized. For each period, the subject will receive one drop in each eye for one day. A 1-4 day washout will separate each period.
  Interventions: Other: FID123300 ocular lubricant; Other: FID123301 ocular lubricant; Other: FID122505 ocular lubricant
- FID122505/FID123300/FID123301 (Other): FID122505 ocular lubricant in Period 1, followed by FID123300 ocular lubricant in Period 2, followed by FID123301 ocular lubricant in Period 3, as randomized. For each period, the subject will receive one drop in each eye for one day. A 1-4 day washout will separate each period.
  Interventions: Other: FID123300 ocular lubricant; Other: FID123301 ocular lubricant; Other: FID122505 ocular lubricant

INTERVENTIONS:
Other: FID123300 ocular lubricant — Investigational ocular lubricant
Other: FID123301 ocular lubricant — Investigational ocular lubricant
Other: FID122505 ocular lubricant — Comparator ocular lubricant

SUMMARY:
The purpose of this study is to evaluate investigational ocular lubricants for their safety and tolerability on subjects with mild to moderate dry eye disease.

DETAILED DESCRIPTION:
Subjects will be expected to attend a screening visit followed by 6 additional study visits. The expected duration of subject participation is approximately 3 weeks. This study will be conducted in Australia.

ELIGIBILITY:
Key Inclusion Criteria:

* Sign an Informed Consent;
* Have dry eye symptoms;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Ocular abnormalities;
* Active ocular infection or inflammation not associated with dry eye;
* History of ocular or intraocular surgery;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) with manifest refraction, at distance | Day 1, each wear period. A wear period is 1 day.
  BCVA will be collected for each eye individually and recorded in logarithm Minimum Angle of Resolution (logMAR)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Dry Eye, Study Director — Alcon Research, LLC
Locations (3):
- Australia (3):
  - George Street Eye Centre, Sydney, New South Wales
  - Ophthalmic Trials Australia, Teneriffe, Queensland
  - University of Melbourne, Department of Optometry and Vision Science, Carlton, Victoria

IPD SHARING:
Plan to Share IPD: No